CLINICAL TRIAL: NCT03675321
Title: Defining Adolescent Nausea Through Brain-Gut Physiology and Non-Invasive Neurostimulation Response
Brief Title: Defining Adolescent Nausea Through Brain Imaging and Neurostimulation Response
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Katja Karrento, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1064187-2; 1K23DK116969-01 (NIH)
Record Dates: First submitted 2018-05-08; First posted 2018-09-18 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Functional Gastrointestinal Disorders
MeSH Terms: conditions — Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, double blind placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants, investigators and study team members blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Auricular Neurostimulation (Experimental): Intervention: Active Percutaneous Electrical Nerve Field Stimulation (PENFS) 5 days/week x 4 weeks
  Interventions: Device: Active Auricular Neurostimulation
- Sham Auricular Neurostimulation (Sham Comparator): Intervention: Sham (Inactive) Percutaneous Electrical Nerve Field Stimulation (PENFS) 5 days/week x 4 weeks.
  Interventions: Device: Sham Auricular Neurostimulation

INTERVENTIONS:
Device: Active Auricular Neurostimulation — Active auricular neurostimulation for 4 weeks. Subjects in Active group who do not have significant improvement after 4 weeks may receive an additional 4 weeks of active neurostimulation therapy.
  Other Names: Percutaneous Electrical Nerve Field Stimulation (PENFS); Neuro-Stim System-2
  Arms: Auricular Neurostimulation
Device: Sham Auricular Neurostimulation — Sham auricular neurostimulation for 4 weeks with identical device as the active but lacking the electrical charge.
  Subjects in Sham group who do not have significant improvement after 4 weeks may receive an additional 4 weeks of active neurostimulation therapy.
  Other Names: Sham neurostimulation without electrical charge
  Arms: Sham Auricular Neurostimulation

SUMMARY:
This study evaluates the efficacy of auricular neurostimulation via an non-invasive percutaneous electrical nerve field stimulator (PENFS) in adolescents with functional nausea. A neurostimulator is applied to the outer ear and stimulates several nerves that are thought to be involved in transmission of nausea and vomiting signals. Half of the study subjects will receive an active nerve stimulator while the other half will receive an inactive one.

DETAILED DESCRIPTION:
By stimulating branches of several cranial nerves in the outer ear, this study aims to improve symptoms and quality of life in adolescents with functional nausea.

The study has the following specific aims:

1. To define adolescent functional nausea into subtypes based on clinical characterization and physiologic testing.
2. Evaluating the efficacy of auricular neurostimulation via PENFS for functional nausea. Subjects will be randomized into two groups: 1) neurostimulation versus 2) sham. They will receive either an active or non-active (sham group) device for 5 days each week x 4 weeks total. Those who do not improve will receive an additional 4 weeks of therapy with active stimulation.
3. Investigate possible brain functional connectivity changes induced by auricular neurostimulation compared to patients with irritable bowel syndrome and healthy controls

ELIGIBILITY:
Inclusion Criteria:

* Meeting pediatric Rome IV criteria for functional nausea
* English-speaking and able to verbalize their condition and concerns about nausea, pain and other symptoms
* Lack of other explanation for symptoms
* Intact external ear that is free of infection or severe dermatological conditions, - - No currently implanted electrical device

Exclusion Criteria:

* Medically complex and/or suffering from medical condition that may explain symptoms
* Taking a medication that may explain symptoms
* Significant developmental delays
* Patients treated with a new drug affecting the central nervous system within 4 weeks of study start
* Infection or severe dermatological condition of ear
* Currently implanted electrical device
* Patients with a history of severe allergy to adhesives

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 109 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katja Kovacic, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Children's Hospital of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babygirija R, Sood M, Kannampalli P, Sengupta JN, Miranda A. Percutaneous electrical nerve field stimulation modulates central pain pathways and attenuates post-inflammatory visceral and somatic hyperalgesia in rats. Neuroscience. 2017 Jul 25;356:11-21. doi: 10.1016/j.neuroscience.2017.05.012. Epub 2017 May 17. PMID 28526575
- [Background] Roberts A, Sithole A, Sedghi M, Walker CA, Quinn TM. Minimal adverse effects profile following implantation of periauricular percutaneous electrical nerve field stimulators: a retrospective cohort study. Med Devices (Auckl). 2016 Nov 3;9:389-393. doi: 10.2147/MDER.S107426. eCollection 2016. PMID 27843360
- [Result] Kovacic K, Hainsworth K, Sood M, Chelimsky G, Unteutsch R, Nugent M, Simpson P, Miranda A. Neurostimulation for abdominal pain-related functional gastrointestinal disorders in adolescents: a randomised, double-blind, sham-controlled trial. Lancet Gastroenterol Hepatol. 2017 Oct;2(10):727-737. doi: 10.1016/S2468-1253(17)30253-4. Epub 2017 Aug 18. PMID 28826627

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: n=1 participant excluded after enrollment but prior to randomization due to ineligibility (alternate diagnosis discovered)
Groups:
- Auricular Neurostimulation: Intervention: Active Percutaneous Electrical Nerve Field Stimulation (PENFS) 5 days/week x 4 weeks
  Active Auricular Neurostimulation: Active auricular neurostimulation for 4 weeks.
  Subjects in Active group who do not have significant improvement after 4 weeks may receive an additional 4 weeks of active neurostimulation therapy.
- Sham Auricular Neurostimulation: Intervention: Sham (Inactive) Percutaneous Electrical Nerve Field Stimulation (PENFS) 5 days/week x 4 weeks.
  Sham Auricular Neurostimulation: Sham auricular neurostimulation for 4 weeks with identical device as the active but lacking the electrical charge.
  Subjects in Sham group who do not have significant improvement after 4 weeks may receive an additional 4 weeks of active neurostimulation therapy.
Period: Overall Study
Arm/Group | Auricular Neurostimulation | Sham Auricular Neurostimulation
Started | 54 | 54
Completed | 51 | 49
Not Completed | 3 | 5
Not completed — Lack of Efficacy | 2 | 2
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: 4 participants excluded from analyses (n=1 treatment and n=3 sham) due to baseline scores of zero on primary outcome (n=3) and alternate diagnosis discovered (n=1)
Groups:
- Total: Total of all reporting groups
Arm/Group | Auricular Neurostimulation | Sham Auricular Neurostimulation | Total
Number analyzed (Participants) | 50 | 46 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 48 | 46 | 94
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 15.04 [13.25 to 16.67] | 15.79 [14.00 to 16.67] | 15.13 [13.33 to 16.67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 38 | 77
  Male | 11 | 8 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 48 | 45 | 93
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 50 | 46 | 96
Nausea Severity Scale [Median (Inter-Quartile Range); unit: units on a scale] — Nausea Severity Scale measures 1) frequency of nausea on a scale 0-4 over past week (0=not at all; 4=every day), 2) average number of nausea episodes/day over past week on a scale 0-4 (0=none; 4=constant), 3) average duration of nausea episodes over past week on scale 0-4 (0=none; 4=most or all of day) and 4) severity of nausea on scale 0-10 (0=none;10=most nausea possible). The severity subscale is converted to a 5 point scale ranging from 0-4. The mean of all 4 subscales yields a total score ranging from 0 to 4, with a higher score indicating more severity.
  units on a scale | 2.85 [2.45 to 3.40] | 2.75 [2.25 to 3.50] | 2.78 [2.28 to 3.43]
Nausea Profile [Median (Inter-Quartile Range); unit: units on a scale] — Nausea Profile measures 3 dimensions of nausea (Emotional, GI and Somatic distress) with 17 items. Each sub scale is measured on a 10-point scale from 0-9 (0=not at all; 9=severely). Total score is calculated as follows: actual score/153 * 100%. Subscales are similarly computed into a percentage score. Higher percentage indicates worse outcomes.
  units on a scale | 44.44 [31.37 to 60.78] | 49.67 [32.03 to 67.32] | 47.08 [32.03 to 62.75]
Baxter Retching faces scale [Median (Inter-Quartile Range); unit: units on a scale] — Baxter Retching faces scale measures daily nausea severity on a pictorial faces scale from 0-10 (0=no nausea; 10=most nausea possible). Weekly averages will be computed and change from baseline to average severity during last week of therapy will be assessed. Higher values indicate worse outcome.
  units on a scale | 2.83 [2.00 to 4.57] | 3.14 [2.00 to 4.00] | 2.99 [2.00 to 4.29]

OUTCOME MEASURES:

1. Primary Outcome: Nausea Severity Scale
Description: Measures 1) frequency of nausea on a scale 0-4 over past week (0=not at all; 4=every day), 2) average number of nausea episodes/day over past week on a scale 0-4 (0=none; 4=constant), 3) average duration of nausea episodes over past week on scale 0-4 (0=none; 4=most or all of day) and 4) severity of nausea on scale 0-10 (0=none;10=most nausea possible). The severity subscale is converted to a 5 point scale ranging from 0-4. The mean of all 4 subscales yields a total score ranging from 0 to 4, with a higher score indicating more severity.
Time Frame: After 4 weeks of therapy
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- Auricular Neurostimulation: Intervention: Active Percutaneous Electrical Nerve Field Stimulation (PENFS) 5 days/week x 4 weeks
  Active Auricular Neurostimulation: Active auricular neurostimulation for 4 weeks.
- Sham Auricular Neurostimulation: Intervention: Sham (Inactive) Percutaneous Electrical Nerve Field Stimulation (PENFS) 5 days/week x 4 weeks.
  Sham Auricular Neurostimulation: Sham auricular neurostimulation for 4 weeks with identical device as the active but lacking the electrical charge.
Arm/Group | Auricular Neurostimulation | Sham Auricular Neurostimulation
Number analyzed (Participants) | 50 | 46
units on a scale | 2.18 [1.55 to 3.30] | 2.45 [1.60 to 3.10]

2. Secondary Outcome: Nausea Profile
Description: Measures 3 dimensions of nausea (Emotional, GI and Somatic distress) with 17 items. Each sub scale is measured on a 10-point scale from 0-9 (0=not at all; 9=severely). Total score is calculated as follows: actual score/153 * 100%. Subscales are similarly computed into a percentage score. Higher percentage indicates worse outcomes.
Time Frame: After 4 weeks of therapy
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Auricular Neurostimulation | Sham Auricular Neurostimulation
Number analyzed (Participants) | 50 | 46
units on a scale | 33.33 [15.69 to 49.02] | 28.43 [16.34 to 51.63]

3. Secondary Outcome: Baxter Retching Faces Scale
Description: Measures daily nausea severity on a pictorial faces scale from 0-10 (0=no nausea; 10=most nausea possible). Weekly averages will be computed and change from baseline to average severity during last week of therapy will be assessed. Higher values indicate worse outcome.
Time Frame: Average score during week 4 of therapy
Population: Some missing data as not all participants completed the daily diaries
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Auricular Neurostimulation | Sham Auricular Neurostimulation
Number analyzed (Participants) | 37 | 33
units on a scale | 2.29 [1.14 to 4.00] | 3.43 [1.67 to 4.86]

ADVERSE EVENTS:
Time Frame: Weekly assessment during intervention and at follow-up visits after end of study for a total of 6 months.
Description: Adverse events assessed by research nurse and research coordinator weekly during treatment intervention and at all follow up visits.
Arm/Group | Auricular Neurostimulation | Sham Auricular Neurostimulation
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/46
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/46
Other Adverse Events (participants affected / at risk) | 11/50 | 16/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Auricular Neurostimulation (N=50) | Sham Auricular Neurostimulation (N=46)
Skin irritation (Skin and subcutaneous tissue disorders) | 5 | 11 — Mild skin irritation from adhesive
Local discomfort (General disorders) | 4 | 4 — Local discomfort at site of electrode placement
Headache (Nervous system disorders) | 1 | 0 — Mild headache, possible related to intervention. Resolved.
Dizziness (Nervous system disorders) | 1 | 0 — mild, possibly related to intervention
Nausea (Gastrointestinal disorders) | 0 | 1 — Moderate; possibly related to intervention

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT03675321/Prot_SAP_000.pdf